CLINICAL TRIAL: NCT04234477
Title: Assessment of Intravenous Rate Control Response in Atrial Fibrillation Trial Pilot Study (AIRCRAFT)
Brief Title: Assessment of Intravenous Rate Control Response in Atrial Fibrillation Trial (AIRCRAFT)
Acronym: AIRCRAFT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was not IRB approved and there were anticipated challenges in recruiting participants.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-39217
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation
Keywords: beta-blocker; calcium channel blocker; rapid ventricular rate (RVR)
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metoprolol; esmolol; Diltiazem; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Beta-blocker strategy (Experimental): MICU patients assigned to Team Blue will receive an intravenous (IV) beta-blocker strategy to manage AF with RVR
  Interventions: Drug: Beta-blocker strategy
- Calcium channel blocker strategy (Experimental): MICU patients assigned to Team Red will receive an intravenous (IV) calcium channel blocker strategy to manage AF with RVR
  Interventions: Drug: Calcium channel blocker strategy
- Physician preference strategy (Active Comparator): MICU patients assigned to Team Green will receive a physician preference strategy with usual/standard of care interventions to manage AF with RVR
  Interventions: Drug: Physician preference strategy

INTERVENTIONS:
Drug: Beta-blocker strategy — Clinicians within the intervention groups will be free to use whatever dosing amount and frequency of their assigned medication class that they deem as medically appropriate, including the decision to use intermittent IV boluses versus continuous infusions.
  Other Names: metoprolol or esmolol
  Arms: Beta-blocker strategy
Drug: Calcium channel blocker strategy — Clinicians within the intervention groups will be free to use whatever dosing amount and frequency of their assigned medication class that they deem as medically appropriate, including the decision to use intermittent IV boluses versus continuous infusions.
  Other Names: diltiazem and verapamil
  Arms: Calcium channel blocker strategy
Drug: Physician preference strategy — This strategy allows for "usual care," with providers selecting their preferred rate-control agent. IV beta-blockers available through the inpatient pharmacy include metoprolol or esmolol, and IV calcium channel blockers include diltiazem and verapamil.
  Arms: Physician preference strategy

SUMMARY:
The Assessment of Intravenous Rate Control Response in Atrial Fibrillation Trial Pilot Study (AIRCRAFT Pilot) is a prospective, unblinded, pragmatic, cluster-level allocation trial. AIRCRAFT compares two medication classes commonly used for rate control in patients in atrial fibrillation (AF) with rapid ventricular rate (RVR). The purpose of this pilot study is to evaluate the feasibility and approach to conducting a trial that compares the use of IV beta blockers and IV calcium channel blockers for patients in AF with RVR in the medical intensive care unit (MICU). AF with RVR is considered when the following parameters are met: (1) Cardiac rhythm consistent with AF (2) Heart rate > 110 bpm. AF with RVR recurrence after conversion to sinus rhythm or prior rate control will count as a new episode of AF with RVR. Rate control agents will be pseudo-randomized to each of the three different MICU teams (beta-blocker, calcium channel blocker and physician preference). Patients are admitted to the three MICU teams on a rotating basis which will allow for pseudo-randomization, the effects of which will be equal between the three teams. Patients will be enrolled in the study if they develop AF with RVR and will be followed until discharge from the MICU. This study aims to assess the adherence and fidelity to treatment assignments in the current novel pilot study protocol which will help inform the feasibility of a larger-scale efficacy trial between IV beta blockers and IV calcium channel blockers for initial management of AF with RVR. Assessment of adherence and fidelity to treatment assignments in management of AF with RVR in the MICU will help inform power calculations and the percent of patients in each study group that received the assigned class of medication will help inform feasibility. Additional aims include assessment of time from medication administration to rate control or sinus conversion as well as identifying optimal means of data extraction (manual vs automated), and incidence of adverse events including hypotension and bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* All adults admitted to the MICU at Boston Medical Center (BMC) during the study period who develop AF with RVR whose treating clinicians decides intravenous (IV) rate control agent is necessary to manage AF with RVR
* Patients readmitted to the MICU during the study period with recurrence of AF with RVR after conversion to sinus rhythm or prior rate control

Exclusion Criteria:

* Pregnancy
* Prisoners
* Allergies to study interventions
* Presentation consistent with acute asthma exacerbation
* Presentation consistent with acute systolic heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Adherence to assigned class of medication | 6 months
  The proportion of patients with AF with RVR that required rate control and were treated with their assigned class of medication. The proportion will be calculated within each group as the number of patients who received their assigned class of medication divided by the total number of patients who received any treatment for rate control of AF with RVR.

SECONDARY OUTCOMES:
Average number of cases of AF with RVR occurring monthly | 6 months
  The total number of cases of AF with RVR will be divided by the total number of MICU patients for each month of the 6 month study.
Percentage of patients who received an IV rate control agent that had AF with RVR | 6 months
  The number of patients who received an IV rate control agent that had AF with RVR will be divided by the total number of patients who had AF with RVR. Telemetry monitoring or EKG results will be used to identify patients with AF and RVR.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Walkey, MD, Study Director — Pulmonary Center Boston Medical Center
Locations (1):
- Boston Medical Center MICU, Boston, Massachusetts, United States